CLINICAL TRIAL: NCT02613650
Title: A Phase 1b Trial of a Combination of mFOLFIRI With MEK162 in Patients With Advanced RAS (HRAS, NRAS, or KRAS) Positive Metastatic Colorectal Cancers
Brief Title: A Trial of mFOLFIRI With MEK162 in Patients With Advanced RAS (HRAS, NRAS, or KRAS) Positive Metastatic Colorectal Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI87144
Record Dates: First submitted 2015-11-12; First posted 2015-11-24 (Estimated); Last update posted 2024-08-09 (Actual); Status verified 2024-03

CONDITIONS: Advanced KRAS Positive Metastatic Colorectal Cancer
MeSH Terms: interventions — binimetinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MEK162 and mFOLFIRI, all patients (Experimental)
  Interventions: Drug: MEK162 and mFOLFIRI

INTERVENTIONS:
Drug: MEK162 and mFOLFIRI — MEK162 in combination with mFOLFIRI in a 14 day cycle
  MEK162 will be given single agent 6 day lead in and then will be given in combination with mFOLFIRI
  mFOLFIRI Administered Day 1 of each cycle Irinotecan 180mg/m2 iv over 90 minutes on day 1 5-fluoruracil 1200mg/m2 continuous infusion for 48 hours (2400mg/m2 in 48 hours)
  Followed by MEK162 - Taken twice daily orally on Days 1-12 of each cycle
  Level -1: mFOLFIRI at 80% + MEK162 30 mg twice daily 1 week on and 1 week off Level 1: mFOLFIRI + MEK162 30 mg twice daily Level 2: mFOLFIRI + MEK162 45 mg twice daily
  Other Names: Binimetinib

SUMMARY:
This is a Phase 1b, open label, dose-finding study to determine the Maximum Tolerated Dose (MTD) of MEK162 in combination with mFOLFIRI, and to evaluate the response rate, clinical benefit rate and additional safety parameters of the treatment combination

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Patients with histologically confirmed RAS (HRAS, NRAS, or KRAS) positive metastatic colorectal cancer.
* Patients must have progressed during or after first-line treatment for metastatic disease with oxaliplatin and fluoropyrimidines based chemotherapy (with failure within six months) or not be a candidate for oxaliplatin (i.e. neuropathy).
* ECOG Performance Status 0-1
* Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines.
* Adequate bone marrow, organ function and laboratory parameters as defined by the protocol
* Adequate cardiac function as defined by the protocol
* Must have recovered from adverse effects of any prior surgery, radiotherapy or other antineoplastic therapy. Alopecia and CTCAE grade 1 peripheral neuropathy is acceptable
* Willingness and ability to comply with all study procedures and able to take oral medications

Dose Expansion Phase Additional Inclusion Criteria

* Patients must be willing to undergo biopsy according to the institute's own guidelines and requirements for such procedures unless deemed unsafe by the investigator
* Patients must have measurable disease as defined by RECIST v1.1 (at least one lesion ≥ 10mm in at least one dimension when assessed by CT or MRI, or a cutaneous lesion with clearly defined margins that measures ≥ 10 mm in at least one dimension)
* Patients must be irinotecan refractory. Patients must have progressed on prior irinotecan therapy but must be able to tolerate standard irinotecan doses.

Exclusion Criteria:

* UGT1A1 *28 homozygous patients
* Previous treatment with any MEK inhibitor
* Treatment with systemic antineoplastic therapy (including unconjugated therapeutic antibodies and toxin immunoconjugates) or any investigational therapy ≤ 4 weeks (<6 weeks for nitrosurea or mitomycin-C, antibodies except for trastuzumab) or ≤ 5-half lives of the investigational therapy prior to starting study treatment, whichever is longer
* Patient received radiotherapy ≤ 2 weeks prior to the first dose of study treatment except localized radiation therapy for symptomatic bone metastasis.
* Have had a diagnosis of another malignancy, unless the patient has been disease-free for at least 3 years following the completion of curative intent therapy, with the following exceptions:

  * Patients with treated non-melanoma skin cancer, in situ carcinoma, or cervical intraepithelial neoplasia, regardless of the disease-free duration, are eligible for this study if definitive treatment for the condition has been completed.
  * Patients with organ-confined prostate cancer with no evidence of recurrent or progressive disease based on prostate-specific antigen (PSA) values are also eligible for this study if hormonal therapy has been initiated or a radical prostatectomy has been performed.
* History or current evidence of retinal vein occlusion (RVO) or current risk factors for RVO (e.g. uncontrolled glaucoma or ocular hypertension, history of hyperviscosity or hypercoagulability syndromes.
* Personal history of Gilbert's syndrome.
* Uncontrolled arterial hypertension defined by blood pressure >150 mmHg systolic and/or 100 mmHg diastolic at rest (average 3 consecutive readings at least 5 minutes apart) despite appropriate medical therapy.
* Impaired cardiovascular function or clinically significant cardiovascular diseases, including any of the following:

  * History of acute coronary syndromes (including myocardial infarction, unstable angina, coronary artery bypass grafting, coronary angioplasty, or stenting) <6 months prior to screening,
  * Symptomatic chronic heart failure; evidence of clinically significant cardiac arrhythmias and/or conduction abnormalities < 6 months prior to screening except atrial fibrillation and paroxysmal supraventricular tachycardia.
* Known positive serology for HIV, active Hepatitis B, and/or active Hepatitis C infection (Note: if not suspected, testing is not required at baseline).
* Patients who have neuromuscular disorders that are associated with elevated CK (e.g., inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis, spinal muscular atrophy).
* Patients who are planning on embarking on a new strenuous exercise regimen after first dose of study treatment. Muscular activities, such as strenuous exercise, that can result in significant increases in plasma CK levels should be avoided while on MEK162 treatment.
* Impairment of gastrointestinal function or gastrointestinal disease (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection that under the judgment of the PI may impair absorption of study drugs).
* Any other condition that would, in the Investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures, e.g., infection/inflammation, intestinal obstruction, unable to swallow medication.(patients may not receive drug through a feeding tube), social/ psychological issues, etc.
* Patients who have undergone major surgery ≤ 3 weeks prior to starting study drug or who have not recovered from side effects of such procedure.
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test.

  * A positive β-hCG result will not be exclusionary if it is suspected to originate from a malignancy and the patient has undergone a confirmatory ultrasound within 72 hours prior to starting MEK162 therapy.
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception from screening through 30 days after the last dose of study drug/treatment discontinuation.
* Sexually active males, unless they use a condom during intercourse while taking the drug through 90 days after the end of systemic exposure to study drug/treatment. In addition, male participants should not father a child in this period and must refrain from donating sperm during the study through 90 days after the end of systemic exposure of study drug/treatment. A condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid.
* Medical, psychiatric, cognitive or other conditions that may compromise the patient's ability to understand the patient information, give informed consent, comply with the study protocol or complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-08-19 (Actual); Primary Completion 2022-11-23 (Actual); Study Completion 2022-12-21 (Actual)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities (DLTs) of combination MEK162 and mFOLFIRI | Patient safety will be evaluated throughout the treatment period (treatment with MEK162 and mFOLFIRI which is expected to last 6-10 months for each patient)

SECONDARY OUTCOMES:
Response Rate | 2 months
  Changes in size of target lesions according to RECIST 1.1 to assess PR/CR
Clinical benefit rate | 4 months
  Changes in size of target lesions according to RECIST 1.1 to assess PR/CR/SD at 4 months
Additional Safety | 9 months
  Incidence of adverse events
Progression-free survival | 9 months

CONTACTS AND LOCATIONS:
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2017-11-02): https://cdn.clinicaltrials.gov/large-docs/50/NCT02613650/Prot_001.pdf